CLINICAL TRIAL: NCT06508775
Title: Long-Term Follow-up of Patients Treated With Miltenyi Cell and Gene Therapies
Acronym: LONGSAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M-2022-393; 2022-501648-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-11; First posted 2024-07-18 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-08

CONDITIONS: Melanoma Stage III; B-cell Non Hodgkin Lymphoma; Pediatric ALL; Childhood Non-Hodgkin Lymphoma; Acute Lymphatic Leukemia; Chronic Lymphatic Leukemia; Melanoma Stage IV
MeSH Terms: conditions — Melanoma; Lymphoma, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: Single dose treatment with CAR T cell therapy in previous trial, long-term follow-up in this trial with cohorts: MB-CART20.1 Lymphoma, MB-CART20.1 Melanoma, MB-CART19.1 pediatric ALL and progressive NHL, MB-CART19.1 adult ALL, MB-CART19.1 adult NHL/CLL, MB-CART2019.1 Lymphoma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long-term follow-up of CAR T cell therapy (Experimental): Assessment of long-term safety and efficacy of Miltenyi CAR T treatment.
  Interventions: Biological: MB-CART19.1; Biological: MB-CART20.1; Biological: MB-CART2019.1

INTERVENTIONS:
Biological: MB-CART19.1 — Assessment of long-term safety and efficacy of MB-CART19.1 treatment.
  Other Names: CD19-targeting CAR T cells; Anti-CD19 CAR T cells
Biological: MB-CART20.1 — Assessment of long-term safety and efficacy of MB-CART20.1 treatment.
  Other Names: CD20-targeting CAR T cells; Anti-CD20 CAR T cells
Biological: MB-CART2019.1 — Assessment of long-term safety and efficacy of MB-CART2019.1 treatment.
  Other Names: CD20/CD19-targeting CAR T cells; Anti-CD20/CD19 CAR T cells

SUMMARY:
The goal of this Long-Term Follow-Up Trial is to assess long-term safety and efficacy of Miltenyi CAR T treatment.

DETAILED DESCRIPTION:
The focus in this trial is on the occurrence of any late adverse reactions (AR), serious adverse events (SAE), serious adverse reactions (SAR) and adverse events of special interest (AESI), i.e. relapse or progression of the underlying disease, life-threatening infections, death due to any case, new and secondary malignancies, lymphocyte counts, detection of the transgene of the CAR T cells, detection of replication-competent lentivirus (RCL), developmental tracking in pediatric patients and furthermore, assessment of the primary status of disease progression and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient underwent treatment with a Miltenyi CAR T cell therapy in one of the parent trials at least 12 months prior to enrollment in long-term follow-up.
* Patient has provided informed consent prior to enrollment.

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | through study completion, up to 14 years
  Percentage of patients with late-onset adverse reactions (AR), serious adverse events (SAE), serious adverse reactions (SAR) and adverse events of special interest (AESI) including relapse or progression of the underlying disease, life-threatening infections, death due to any cause, new and secondary malignancies

SECONDARY OUTCOMES:
Lymphocyte count | through study completion, up to 14 years
  B and T lymphocyte count
Height | through study completion, up to 14 years
  Height
Weight | through study completion, up to 14 years
  Weight
Tanner staging for pediatric patients | through study completion, up to 14 years
  Tanner staging for pediatric patients
Menstruation status for pediatric patients | through study completion, up to 14 years
  Did the patient experience their first menstrual cycle (menarche)? If yes, enter date
RCL | through study completion, up to 14 years
  Percentage of patients with detectable replication-competent lentivirus (RCL) (if results of 2 consecutive years are negative for an individual patient, further sampling will not be continued for this patient; if results of all samples in first year of primary trial were negative for an individual patient, sampling will not be continued for this patient in this long-term follow-up trial)
Relapse / Progression | through study completion, up to 14 years
  Percentage of patients who relapse or progress since enrollment and rate of surviving patients
Detectable Transgene levels | through study completion, up to 14 years
  Percentage of patients with detectable transgene levels (if results of 2 consecutive years are negative for an individual patient, further sampling will be stopped for this patient)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Rössig, Prof. Dr., Principal Investigator — Universitätsklinikum Münster
Locations (7):
- Germany (7):
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Köln, Cologne
  - Uniklinikum Erlangen, Erlangen
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen
  - Universitäts-Kinderklinik Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No